CLINICAL TRIAL: NCT00366769
Title: Evaluation of Visual Outcomes, Contrast Sensitivity, Glare, and Induction of High Order Aberrations Following LASIK Surgery Using CustomVue
Brief Title: Evaluation of Outcomes Following LASIK Surgery Using CustomVue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRC-05-005
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2006-08-21 (Estimated); Status verified 2006-03

CONDITIONS: Myopia; Astigmatism; Myopic Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

INTERVENTIONS:
Device: Wavefront-guided LASIK using CustomVue platform

SUMMARY:
The aim of the study was to evaluate visual outcomes, contrast sensitivity, glare and induced high order aberrations induced by the new CustomVue software use for wavefront-guided LASIK.

ELIGIBILITY:
Inclusion Criteria:

* Myopia 0.00 to -6.00 D
* Astigmatism 0.00 up to -3.00 D
* Manifest refraction spherical equivalent (MRSE) up to -6.00 D.

Exclusion Criteria:

* History of ocular pathology
* Previous ocular surgery
* Large pupils (greater than 8mm diameter, infrared measurement)
* Thin corneas (preoperatively calculated minimal residual bed < 250 um)
* Irregular astigmatism
* Asymmetric astigmatism
* Unstable refraction
* Any other condition that precludes the patient from undergoing LASIK

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-09; Study Completion 2006-02

PRIMARY OUTCOMES:
Visual acuity
Induction of high order aberrations

SECONDARY OUTCOMES:
Contrast sensitivity & glare
Patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Kerry D. Solomon, MD, Principal Investigator — Medical University of South Carolina